CLINICAL TRIAL: NCT00564135
Title: Postoperative Urinary Retention and UTI After LAVH for Benign Disease
Brief Title: Postoperative Urinary Retention and Urinary Track Infection (UTI) After Laparoscopic Assisted Vaginal Hysterectomy (LAVH) for Benign Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Obstetrics and Gynecology, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96-0424C
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2008-08

CONDITIONS: Hysterectomy; Urinary Retention; Urinary Tract Infection
Keywords: hysterectomy; laparoscopy; urinary retention; urinary tract infection; catheterization
MeSH Terms: conditions — Urinary Retention; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A B C (Experimental): A-no Foley B-remove Foley at 7AM in the morning of postoperative day 1 C-remove Foley at 7AM in the morning of postoperative day 2
  Interventions: Procedure: on Foley time

INTERVENTIONS:
Procedure: on Foley time — A-no Foley B-remove Foley at 7AM in the morning of postoperative day 1 C-remove Foley at 7AM in the morning of postoperative day 2

SUMMARY:
With the advent of minimally invasive surgery, laparoscopic assisted vaginal hysterectomy (LAVH) is currently advocated as an alternative to abdominal hysterectomy. Reported benefits of LAVH in short-term study, when compared with the abdominal hysterectomy, include shorter hospital stays and convalescence, less postoperative pain, lower morbidity. To our best knowledge, no study has been conducted to examine bladder catheterization is associated with PUR and UTI after LAVH. No study has been performed to evaluate the long-term sequelae of PUR after LAVH.

In this study, 150 patients undergoing LAVH are randomly assigned to have an indwelling Foley catheter for 0 (n = 50), at 7AM-8AM in the morning of postoperative day 1 (n = 50), at 7AM-8AM in the morning of postoperative day 2 (n = 50) after the procedure by selecting a sealed envelope, which is opened before the operation. The inclusion criteria are uterine fibroids, endometriosis, abnormal bleeding, uterine prolapse and intra-epithelial neoplasia of the cervix grade 3. Patients are excluded if they experienced pelvic reconstructive surgery for pelvic organ prolapse or stress urinary incontinence; if they have bacteriuria and clinical urinary tract symptoms, e.g. dysuria, frequency, urgency and stress incontinence before surgery. After surgery, all patients stay at least 2 days in the hospital. The incidences of febrile morbidity and other postoperative complications are recorded. The outcome is assessed as immediate postoperative urinary tract symptoms, urinary tract bacteriuria (defined as a positive culture > 105 organisms/µl), postoperative fever > 38°C and urinary retention or the inability to pass urine 6 hours after catheter remove. All patients are followed up at 3 months and one year after surgery. To demonstrate quality of life of women after undergo LAVH, a generic instrument of MOS Short Form 36 (SF-36) and two specific instruments for urinary problems, Incontinence Impact Questionnaire (IIQ7) and Urinary Distress Inventory (UDI) are asked to answer in all patients before surgery and postoperative follow-up. All data are analyzed by the two-tailed Fisher exact test when appropriate. Correlation coefficients are calculated to determine the associations of preoperative, intraoperative, and postoperative factors with the incidence of postoperative urinary retention and positive urine cultures. A value of p < 0.05 is considered statistically significant.

DETAILED DESCRIPTION:
Hysterectomy is the most common major gynecological operation performed; in previous study, 20% of women will have undergone a hysterectomy by the age of 50 years, mostly for nonmalignant conditions such as uterine fibroids, endometriosis, abnormal bleeding, uterine prolapse and intra-epithelial neoplasia of the cervix grade 3. (1) Fever is the most common perioperative complication of hysterectomy, arising in about 25%. (2) The other early complications associated with hysterectomy including hemorrhage, infection, and injury to adjacent organs, femoral neuropathy, and thromboembolic disease. (3) However, whether hysterectomy is linked to the development of urinary symptoms remains controversial. Some groups observed no effect or improved urinary dysfunction after hysterectomy, (4-7) others reported that hysterectomy is the cause of a variety of urinary symptoms including the urethral syndrome, stress incontinence, detrusor overactivity and voiding difficulty. (8, 9) Voiding difficulty in the female is a condition in which the bladder fails to empty completely and easily after micturition. Failure to detect voiding difficulties after surgery may lead to bladder overdistention and irreversible damage of the detrusor muscle. (10) Postoperative urinary retention (PUR) is defined as the inability to void with a full bladder during the postoperative period. The etiology of PUR involves a combination of many factors, including sedation, type of anesthesia, increased sympathetic stimulation, overdistension of bladder by large quantities of fluids given intravenously, pain and anxiety. (11) In the literature, incidence of postoperative urinary retention (PUR) has ranged from 3.8% to 80%, depending on the definition used and the type of surgery performed. (12-15) There is no consensus on how to diagnose PUR and various criteria, such as clinical symptoms, bladder palpation and a fixed time interval or drainage by catheterization of more than 500 ml of urine, have been used. (16) Traditionally gynecologists have used an indwelling catheter for abdominal surgical procedures for several reasons, including the beliefs that women would be unable to void satisfactorily in the immediate postoperative period, that the indwelling catheter provided the only reliable method of assuring adequate exposure, and that a catheter would be necessary in the recording of intake-output. In fact, prompted by women's dislike of the catheter as well as an increased incidence of postoperative urinary tract infection (UTI). (17) The potential sequelae of UTI include gram-negative bacteremia, antimicrobial toxicity, chronic bacteriuria and chronic renal disease. (18) In most cases the infection is mild and easily treated, but UTI is the commonest nosocomial infection and leads to increased morbidity and treatment costs. (18-20) Some North American studies addressing postoperative UTI have been confounded by the use of perioperative antibiotics, (17, 21) suggesting UTI rates of 3-10%, whereas British work has suggested a rate of 35% in control patients receiving no antibiotics. (22) It has been estimated that the risk of UTI associated with indwelling catheterization is 5-10% per day of catheterization (18) and that the commonest cause of UTI in hospital is urinary catheterization (23). Short-term catheterization has been associated with subsequent bacterial colony counts of > 105/ml of urine in 21% of women undergoing minor surgery, (24) and the incidence of positive urine cultures rises with the length of time catheterization is continued. (17, 18) In a randomized trial study for the effect of prophylactic antibiotics on the postoperative UTI in patients undergoing abdominal hysterectomy, Ireland et al found single dose cotrimoxazole is effective in reducing the incidence of postoperative UTI from 35% in the control group to 4% in the treated group. (25) Hakvoort et al studied whether prolonged urinary bladder catheterization after vaginal prolapse surgery is advantageous. (26) They found that residual volumes > 200 ml and need for recatheterization occurred in 9% in the 4 days catheterization group versus 40% of patients in the one day catheterization group (OR 0.15, 95% CI 0.045-0.47). Positive urine cultures were found in 40% of cases in the 4 days catheterization group versus 4% of patients in the one day catheterization group (OR 15, 95% CI 3.2-68.6). By contrast, in a prospective study of postoperative infection after abdominal and vaginal gynecological surgery, Kingdom et al reported 40% of 115 patients receiving no prophylactic antibiotics developed a UTI in the postoperative period and this was not clearly related to the need for postoperative catheterization. (25) Since prolonged indwelling urinary catheterization may be associated with an increased risk of UTI, increasing patient morbidity and potentially prolonging the hospital stay (18), prophylactic antibiotics and a reduction in catheter time or no catheter after surgery might be expected to reduce this risk.

Regarding the relationship of bladder catheterization with PUR, in published data of prospective or retrospective studies on PUR after abdominal or vaginal hysterectomy, we found that several factors of postoperative care affect the result of PUR including type of surgery, use of catheter, duration of catheterization, and postoperative analgesia. (16, 17, 25, 27-30) During 4-year period, Summitt et al have not used postoperative bladder catheter drainage after routine vaginal hysterectomy. (28) To assess the potential differences in postoperative outcome, they prospectively compared the use of indwelling bladder catheter drainage with no catheter use after standard vaginal hysterectomy. Their data showed 2 patients in the catheterized group required recatheterization after the catheters were removed; none in the no-catheter group required a catheter. The results inferred that indwelling catheterization appears unnecessary after routine vaginal hysterectomy. In a prospective randomized trial study, Dobbs et al compared the infection rate and postoperative morbidity between indwelling catheterization and in-out catheterization at the time of abdominal hysterectomy. (27) Of the 95 patients in their study, 36% of that undergoing in-out catheterization had PUR, requiring bladder emptying, compared with 4% of those receiving an indwelling catheter. In addition, 29% of the catheterized group had urinary tract bacteriuria compared with 13% of the uncatheterized group. They concluded that in-out urinary catheterization at the time of routine abdominal hysterectomy was associated with a significantly higher incidence of PUR compared with indwelling catheterization, and may have implications for long-term bladder function. (27) Dobbs et al also pointed out that abdominal muscular pain when the intra-abdominal pressure is increased during voiding coupled with the decreased sensation for voiding due to analgesia, suggests that an indwelling catheter in the immediate postoperative period will help to prevent long-term morbidity from bladder atony. Bodker and Lose presented the prevalence of PUR was 9.2% in their patients receiving gynecological surgery. (16) Of 124 patients undergoing abdominal hysterectomy, 13.7% had PUR. Of 24 patients undergoing laparoscopic assisted vaginal hysterectomy (LAVH), 8.7% had PUR. They concluded patients at risk of PUR are difficult to predict. The risk is higher after laparotomy than after laparoscopy. A retention rate of 13.7% after abdominal hysterectomy is fairly similar to that of 11.8% after gynecologic laparotomies reported by Schiotz, (29) Who used an indwelling Foley catheter routinely for 20-24 hours to ascertain the risks of UTI and aymptomatic bacteriuria. Based on 949 gynecologic laparotomies without the use of catheters but with bladder needling at the end of surgery, Bartzen and Halferty found that 26% needed catheterization. (17) They suggested that abstaining from the use of an indwelling catheter was also associated with lower cost and greater patient satisfaction.

With the advent of minimally invasive surgery, LAVH is currently advocated as an alternative to abdominal hysterectomy. Reported benefits of LAVH in short-term study, when compared with the abdominal hysterectomy, include shorter hospital stays and convalescence, less postoperative pain, lower morbidity, and, in some series, greater cost-effectiveness. (31-35) Whereas benefits of LAVH in long-term follow-up, only few studies have appeared in the literature. A report from Taiwan, Shen et al compared 1-month and 8-year follow-up of LAVH and abdominal hysterectomy. In their 8-year follow-up showed no statistically significant differences in vaginal vault prolapse, cystocele, rectocele, enterocele, postcoital bleeding, and cuff granulation between LAVH and abdominal hysterectomy procedures. (36) However, with regard to the consequences of PUR and UTI after LAVH, to our best knowledge, no study has been conducted to examine bladder catheterization is associated with this problem. Furthermore, no study has been performed to evaluate the long-term sequelae of PUR after LAVH.

ELIGIBILITY:
Inclusion Criteria:

* Uterine fibroids
* Endometriosis
* Abnormal bleeding
* Uterine prolapse and intra-epithelial neoplasia of the cervix grade 3

Exclusion Criteria:

* If they experienced pelvic reconstructive surgery for pelvic organ prolapse or stress urinary incontinence
* If they have bacteriuria and clinical urinary tract symptoms, e.g. dysuria, frequency, urgency and stress incontinence before surgery

Ages: 34 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chung Liang, MA, Principal Investigator — CGMH

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246